CLINICAL TRIAL: NCT04787744
Title: Veterans Affairs Seamless Phase II/III Randomized Trial of STAndard Systemic theRapy With or Without PET-directed Local Therapy for OligoRecurrenT Prostate Cancer (VA STARPORT)
Brief Title: Veterans Affairs Seamless Phase II/III Randomized Trial of STAndard Systemic theRapy With or Without PET-directed Local Therapy for Oligometastatic pRosTate Cancer
Acronym: VA STARPORT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCA-026-20S; CX002277-01 (Other Grant/Funding Number: VA Clinical Science Research & Development)
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer; Oligometastasis; Oligorecurrence; Recurrent Prostate Cancer; Metastatic Prostate Cancer; De Novo Prostate Cancer
Keywords: Prostate Cancer; Metastasis; Oligorecurrence; PET-directed local therapy; Standard Systemic Therapy; SBRT; Oligometastasis; Oligorecurrent; Metastasis-directed therapy; Salvage Local Therapy; Recurrent Prostate Cancer; Fluciclovine; PSMA; Choline
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Goserelin; histrelin; Leuprolide; Triptorelin Pamoate; Androgen Antagonists; nilutamide; Flutamide; bicalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; relugolix; abiraterone; Prednisone; Methylprednisolone; apalutamide; enzalutamide

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, multi-center seamless phase II to phase III randomized clinical trial designed to compare SST with or without PET-directed local therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Systemic Therapy (SST) (Active Comparator): All Veterans will receive SST (if De novo, Veterans will receive prostate-directed radiation).
  Interventions: Drug: Goserelin, Histrelin, Leuprolide & Triptorelin; Drug: ADT + Nilutamide, Flutamide, & Bicalutamide; Drug: Degarelix & Relugolix; Drug: ADT + Docetaxel +/- prednisone; Drug: ADT + Abiraterone + Prednisone; Drug: ADT + Abiraterone + Methylprednisolone; Drug: ADT + Apalutamide; Drug: ADT + Enzalutamide; Radiation: Prostate-directed Radiation for De novo oligometastatic prostate cancer
- SST + PET-directed local therapy (Experimental): In addition to SST, all Veterans will receive PET-directed local therapy to all metastases using surgery or radiation. If De novo, Veterans will also receive prostate-directed radiation or radical prostatectomy to treat the prostate/prostate bed. The best course of treatment will be determined using shared decision-making between the physician and Veteran.
  Interventions: Procedure: PET-directed Local Therapy using Surgery; Radiation: PET-directed Local Therapy using Radiation; Other: Salvage Local Therapy for locally recurrent disease; Drug: Goserelin, Histrelin, Leuprolide & Triptorelin; Drug: ADT + Nilutamide, Flutamide, & Bicalutamide; Drug: Degarelix & Relugolix; Drug: ADT + Docetaxel +/- prednisone; Drug: ADT + Abiraterone + Prednisone; Drug: ADT + Abiraterone + Methylprednisolone; Drug: ADT + Apalutamide; Drug: ADT + Enzalutamide; Radiation: Prostate-directed Radiation for De novo oligometastatic prostate cancer

INTERVENTIONS:
Procedure: PET-directed Local Therapy using Surgery — Surgery will be used to treat metastases.
  Arms: SST + PET-directed local therapy
Radiation: PET-directed Local Therapy using Radiation — Radiation therapy will be used to treat metastases.
  Radiation options include:
  1. Stereotactic body radiotherapy (SBRT) using 1-10 fractions
  2. Conventionally fractionated radiotherapy using elective nodal radiotherapy and a simultaneous integrated boost to involved nodes
  The selection of the form of metastasis-directed radiotherapy for each metastasis will be determined using shared decision-making between the treating physician and the Veteran.
  Arms: SST + PET-directed local therapy
Other: Salvage Local Therapy for locally recurrent disease — For Veterans who have a local recurrence in addition to oligorecurrent metastatic lesions, they will undergo salvage local therapy using brachytherapy, SBRT, surgery, cryotherapy or HIFU. The selection of modality of salvage local therapy will be determined using shared decision-making between the treating physician and Veteran.
  Arms: SST + PET-directed local therapy
Drug: Goserelin, Histrelin, Leuprolide & Triptorelin — Androgen deprivation therapy (ADT) using an LHRH agonist
Drug: ADT + Nilutamide, Flutamide, & Bicalutamide — ADT adding anti-androgen therapy to an LHRH agonist
Drug: Degarelix & Relugolix — ADT using an LHRH Antagonist.
Drug: ADT + Docetaxel +/- prednisone — Enhanced SST using chemohormonal therapy
Drug: ADT + Abiraterone + Prednisone — Enhanced SST using Abiraterone + Prednisone
Drug: ADT + Abiraterone + Methylprednisolone — Enhanced SST using Abiraterone + Methylprednisolone
Drug: ADT + Apalutamide — Enhanced SST using ADT + Apalutamide
Drug: ADT + Enzalutamide — Enhanced SST using ADT + Enzalutamide
Radiation: Prostate-directed Radiation for De novo oligometastatic prostate cancer — Veterans in ARM 1 will receive prostate-directed RT only and NO treatment to any nodal or distant metastatic sites.
  Acceptable dose/fractionations include 55 Gy in 20 fractions and 36 Gy in 6 fractions.
  Veterans in ARM 2 should receive prostate-directed local therapy using radiotherapy or radical prostatectomy in addition to PET-directed local therapy to metastases.

SUMMARY:
This is a prospective, open-label, multi-center seamless phase II to phase III randomized clinical trial designed to compare SST with or without PET-directed local therapy in improving the castration-resistant prostate cancer-free survival (CRPC-free survival) for Veterans with oligometastatic prostate cancer. Oligometastasis will be defined as 1-10 sites of metastatic disease based on the clinical determination of the LSI which incorporates all imaging, clinical, and pathologic data available.

DETAILED DESCRIPTION:
Prostate Cancer is the most commonly diagnosed cancer among Veterans, comprising 30% of new cancer diagnoses in the VA. Eighty-five percent of men present with localized prostate cancer, which is typically treated with active surveillance or curative local therapy using surgery or radiation therapy. Unfortunately, twenty percent of Veterans undergoing curative local therapy will develop metastatic recurrence. These men typically receive palliative systemic hormonal therapy to control their disease. Despite this, over half of men will have cancer progression within 1-2 years and half will die within 5 years.

Two diverging paradigms have been studied in recent years to improve the survival of men with recurrent metastatic prostate cancer. First, a subset of patients has oligometastatic disease. These patients are hypothesized to have an intermediate clinical state in which ablative local therapy with surgery or radiation to all metastatic sites of disease (metastasis-directed therapy; MDT) can lead to durable disease control and potentially cure in select patients. Recent Phase II randomized trials have demonstrated improved long-term progression-free survival with MDT in the absence of systemic therapy.

Yet, 75% of patients receiving MDT for oligometastatic cancer develop progression in new areas, arguing that systemic therapy is needed to treat occult metastases. This is supported by data demonstrating that earlier palliative hormonal therapy is associated with improved survival. In fact, the second approach that has been studied in recent years, is whether escalating hormonal therapy by adding novel androgen receptor axis targeted agents or chemotherapy improves outcomes in men with metastatic prostate cancer. Multiple phase III randomized trials demonstrate that escalating hormonal therapy with these novel therapeutic agents improves progression-free survival and overall survival dramatically. Therefore, these agents have been integrated as an option into today's standard systemic therapy (SST) for metastatic prostate cancer.

Given the promise of MDT to induce long-term cancer control and the effectiveness of SST to prevent further cancer progression, there is an urgent need to determine whether adding MDT to SST improves disease outcomes further. Additionally, prior studies have excluded patients with local recurrence. However, these comprise a large proportion of Veterans with recurrent oligometastatic prostate cancer. The primary goal of our study is to determine if adding PET-directed local therapy (MDT and treatment of primary tumor [de novo] or primary tumor local recurrence on PET/CT if applicable) improves disease control compared to SST alone in Veterans with oligometastatic prostate cancer. This is a multi-institutional phase II/III randomized trial comparing SST with or without PET-directed local therapy. Other goals of the study are to determine any differences in patterns of cancer progression, survival, and quality of life. We also will determine if certain mutations present in tumor DNA can predict if Veterans will benefit from PET-directed local therapy.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years. Ability to provide Informed Consent for participation in the study ECOG Performance Status 2 at time of enrollment. Prostate cancer, confirmed histologically or cytologically. If original documentation of histology and cytology are not available, documentation of prostate cancer satisfies these criteria. If recurrent, prior curative-intent local therapy to all sites of prostate cancer with either upfront radiotherapy or prostatectomy with or without post-operative radiotherapy.

If recurrent, PSA suspicious for biochemical recurrence after local therapy, with lab value(s) taken prior to start of SST (if current SST has already started) or within 90 days prior to enrollment if not already on SST, and meeting one of the three below categories:

PSA 0.2 ng/ml x 2 after prostatectomy +/- post-operative radiotherapy; Elevation of PSA 2 ng/ml above the nadir after definitive radiotherapy; Or Two consecutively elevated PSAs with evidence of metastasis on the imaging Studies.

-Serum testosterone obtained prior to randomization based on one of the criteria below:

For patients who have a history of a prior episode of therapy with SST agents for prostate cancer, a total testosterone 100 ng/dl after completion of the prior episode of SST and before the start of current SST or within 30 days of starting current SST if the patient has already started SST for recurrence.

For patients who have no prior history of an episode of therapy with SST agents and have already started SST for recurrence, this pre-SST testosterone is not required.

CT or MRI abdomen/pelvis performed prior to start of SST (if current SST has already started) or within 90 days prior to enrollment if not already on SST. The results from the CT component of the PET/CT can be used to fulfill this criterion. This is optional for patients who have a PSMA PET/CT. Yechnetium (Tc99m-MDP) or sodium fluoride (NaF) bone scan (sodium fluoride preferred) performed prior to start of SST (if current SST has already started), or within 90 days prior to enrollment if not already on SST. This is optional for patients who have a PSMA PET/CT. Prostate PET/CT (currently PSMA, Fluciclovine, choline) performed prior to start of SST (if current SST has already started), or within 90 days prior to enrollment if not already on SST.

1-10 lesions suspicious for nodal recurrence or metastasis from prostate cancer as determined by the investigator based on the above imaging studies.

Has already undergone NPOP sequencing or a plan is in place for NPOP sequencing for prostate cancer.

For participants on SST at the time of enrollment only:

Has been on SST for 180 days. For participants with local recurrence after curative-intent local therapy on imaging :

Patients with local recurrence in the prostate, SV, or prostate bed are eligible as long as there is at least 1 nodal or distant metastatic recurrence. Biopsy must confirm local recurrence for patients who have had prior curative-intent radiation to the prostate, SV, or prostate bed.

Candidate for salvage local therapy (refer to Section 10.4) as determined by a urologist or radiation oncologist (depending on the respective modality to be used to treat the local recurrence).

For participants with de novo prostate cancer:

Candidate for prostate-directed radiation.

Exclusion Criteria:

* Any current or prior evidence of castration-resistant prostate cancer, defined as two consecutive rises in serum PSA, obtained at a minimum of 1-week interval, with the final PSA value >/= 1 ng/ml, while having a total testosterone < 50 ng/dl).
* Prior malignancy, except the following:

  * Adequately treated non-melanomatous skin cancer;
  * Adequately treated Stage 0, I, or II cancer from which the patient is currently in complete remission; or
  * Any other cancer from which the patient has been disease free for three years.
* Presence of a symptomatic metastasis that requires palliative radiotherapy.
* Any known brain metastases, presence of leptomeningeal disease, malignant spinal cord compression, or malignant cauda equina syndrome.
* Prior nodal, bone, or visceral metastasis after curative-intent therapy other than those identified on the enrollment imaging studies which make the patient ineligible for PET-directed local therapy (per investigator discretion).
* Prior radiation therapy to any sites requiring PET-directed local therapy or salvage local therapy that will lead to prohibitively high risk of toxicity from subsequent local therapy, as determined by the treating radiation oncologist (if radiation is intended as the study local therapy) or surgeon/urologist (if surgery is intended as the study local therapy).
* Any other previous or current condition, which, in the judgement of the LSI, is likely to interfere with any STARPORT treatments or assessments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with prostate cancer.
Enrollment: 464 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Castration-resistant prostate cancer-free survival (CRPC-free survival) | 4 years
  CRPC-free survival is a time-to-event outcome defined as the length of time from randomization to the first occurrence of failure. The following are forms of failure in the setting of a castrate testosterone level: PSA progression, radiographic progression, symptomatic skeletal event due to progression, and death.

SECONDARY OUTCOMES:
Radiographic progression-free survival (rPFS) | 4 years
  rPFS is a time-to-event outcome defined as the length of time from randomization to radiographic progression of prostate cancer or death.
Clinical progression-free survival (cPFS) | 4 years
  cPFS is a time-to-event outcome defined as the length of time from randomization to radiographic progression on conventional imaging, symptomatic skeletal event due to progression, or death.
Freedom from index lesion progression (FFILP) | 4 years
  FFILP is a time-to-event outcome defined as the length of time from randomization to progression of any of the enrollment index oligorecurrent lesions.
New metastasis-free survival (MFS) | 4 years
  New MFS is a time-to-event outcome (MFS) defined as the length of time from randomization to the development of a new metastasis that was not present at the time of enrollment, or death.
Prostate cancer-specific survival (PCSS) | 4 years
  PCSS is a time-to-event outcome defined as the length of time from randomization to death from prostate cancer.
Overall survival (OS) | 4 years
  OS is a time-to-event outcome defined as the length of time from randomization to death from any cause.
Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 toxicity | 4 years
  Toxicities will be evaluated based on system organ class and a higher number in the grading system is reflective of more severe toxicity.
Patient-reported quality of life measured by the EORTC QLQ-C30 3.0 | 2 years
  The QLQ-C30 is composed of 30 items. These include five functional scales, three symptom scales, a global health status/QoL scale, and six single items. Raw scores will be converted to standardized scores ranging from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Expanded Prostate cancer Index Composite Short Form (EPIC-26) | 2 years
  EPIC-26 contains 26 items in 5 domains (Urinary Incontinence, Urinary Irritative/Obstructive, Bowel, Sexual, and Hormonal). Raw scores are transformed linearly to a 0-100 scale, with higher scores representing better HRQOL.
Patient-reported health-related quality of life measured by the EQ5D-5L | 2 years
  EQ5D-5l consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and each dimension has 5 levels. The digits for the 5 dimensions is combined to describe the health state (higher total reflect a higher health state). There is also a vertical visual analogue scale to be used as a quantitative measure that reflects the patient's own judgement with the endpoints labelled as "The best health you can imagine" and "The worst health you can imagine."

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Solanki, MD MS, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (20):
- United States (20):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - East Orange Campus of the VA New Jersey Health Care System, East Orange, NJ, East Orange, New Jersey
  - VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, VA, Richmond, Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No